CLINICAL TRIAL: NCT03062631
Title: Treatment Use of 3,4 Diaminopyridine in Congenital Myasthenia
Status: No longer available | Type: Expanded Access
Sponsor: Ricardo Maselli (Other)
Collaborators: Catalyst Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Ricardo Maselli, Professor, University of California, Davis
Organization: University of California, Davis (Other)
Other Study IDs: 223019
Record Dates: First submitted 2017-02-21; First posted 2017-02-23 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Congenital Myasthenic Syndrome
Keywords: Congenital Myasthenic Syndrome; 3,4 DAP; 3,4 Diaminopyridine
MeSH Terms: conditions — Myasthenic Syndromes, Congenital | interventions — Amifampridine

STUDY DESIGN:
Expanded Access Types: Individual, Treatment

INTERVENTIONS:
Drug: 3,4-Diaminopyridine — The investigator will prescribe an initial dose of 3,4 diaminopyridine (DAP) by mouth based on the participant's weight. This initial dose may be modified later according to the participant's response to treatment.
  Other Names: 3,4-DAP

SUMMARY:
Congenital myasthenia is a potentially lethal disorder, which, even with careful management, significantly impedes participation in normal daily functions. Currently approved therapies have had little impact on promoting a normal quality of life activity in these patients. The goal is to systematically examine the effect of 3,4-DAP on the natural course of this disease and to gain additional experience in titrating 3,4-DAP with other available therapies to maximize clinical function and development in this patient population.

The specific aim of this study is to evaluate the use of 3,4 Diaminopyridine (DAP) on selected patients proven by genetic or serum antibody testing to have Congenital Myasthenic Syndrome (CMS), prescribe 3,4 DAP, and then clinically evaluate the response.

DETAILED DESCRIPTION:
The subject population will consist of selected patients proven by genetic testing, muscle biopsy or antibody testing to have CMS. Consideration for entry in our clinical study will require referral from a treating pediatrician or neurologist. Dr. Maselli will examine patients and deem which are appropriate for neurophysiologic examinations at the University of California, Davis Medical Center. In vitro neuromuscular recordings of anconeus muscle biopsy material (as well as standard light and electron morphologic analysis) or documentation of a genetic mutation associated with congenital myasthenia will be required in some patients to confirm the diagnosis of CMS.

If a participant decides to volunteer, and if the diagnosis of Congenital Myasthenic Syndrome (CMS) has not been established, the participant may need to undergo a muscle biopsy or a blood sampling for DNA testing. The investigators will obtain a blood test (serum chemistry) before participants start treatment and then once a year after the start of 3,4-DAP treatment. Participants will also have an electrocardiograph (EKG) before starting treatment, and every 2 years after the start of 3,4-DAP treatment. All study participants will then return to the clinic once each year (or more often if the neurologist feels it is necessary) for follow-up care.

Participants will receive treatment with the study drug until it is approved by the FDA for use in patients with CMS, until the investigator stops the study drug (because it doesn't work for the participant or it is unsafe for to take), or until the study is ended for other reasons (i.e. safety concerns are discovered, etc.), whichever comes first. Participants will be allowed to stay on other medications for myasthenia or add other medications to treat their condition, as necessary.

If participants have an unclear history of episodes resembling seizures as determined by the investigator, they should not to drive or operate heavy machinery for the first 6 months of the study.

Participants may not participate in this study if they are pregnant or breastfeeding or if they are a woman of childbearing potential who plans to become pregnant while on the study. It is unclear how 3,4 DAP can effect an unborn fetus. Therefore, women of childbearing potential will have a pregnancy test prior to starting the study drug and periodically throughout the study, if needed. Participants who think they may have become pregnant during the study should tell the study doctor immediately.

ELIGIBILITY:
Inclusion Criteria:

1. Proven by genetic testing, muscle biopsy or antibody testing to have CMS.
2. Age of 3 months - 75 years old.
3. Willing to take a pregnancy test if female and of child-bearing age.
4. Available for the minimum time commitment (annual visit) required for the study.

Exclusion Criteria:

1. Pregnancy
2. History of allergic reactions to pyridines
3. History of confirmed seizures in the opinion of the study investigator, liver disease, or cardiac arrhythmias. Subjects with a questionable history of episodes that are not clearly seizures as determined by the investigator may participate.

Ages: 3 Months to 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Maselli, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Medical Center, Sacramento, California, United States